CLINICAL TRIAL: NCT01663532
Title: A 12-week, Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Aripiprazole Intramuscular Depot (OPC-14597, Lu AF41155) in the Acute Treatment of Adults With Schizophrenia
Brief Title: Trial of Aripiprazole Intramuscular Depot (OPC-14597, Lu AF41155) in the Acute Treatment of Adults With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry); Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31-12-291
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole IM Depot (Experimental): Aripiprazole IM Depot 400 mg, with allowed decrease to 300 mg for safety and return to 400 mg for efficacy if needed, every four weeks for 12 weeks
  Interventions: Drug: Aripiprazole IM Depot
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole IM Depot
  Other Names: OPC-14597; Lu AF41155
  Arms: Aripiprazole IM Depot
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the overall efficacy of aripiprazole intramuscular (IM) depot as acute treatment in subjects with schizophrenia.

The secondary purpose is to evaluate the safety and tolerability of aripiprazole IM depot administered every 4 weeks for 12 weeks to adult subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 65 years of age, inclusive, at time of informed consent.
* Subjects with a diagnosis of schizophrenia for at least 1 year as defined by DSM-IV-TR criteria and confirmed by the MINI for Schizophrenia and Psychotic Disorders Studies.
* Subjects with a stable living environment when not in hospital.
* Subjects who would benefit from hospitalization or continued hospitalization for treatment of a current acute relapse of schizophrenia at trial entry.
* Subjects who are experiencing an acute exacerbation of psychotic symptoms and marked deterioration of usual function as demonstrated by meeting BOTH of the following at screening and baseline:

  * Currently experiencing an acute exacerbation of psychotic symptoms accompanied by significant deterioration in the subject's clinical and/or functional status from their baseline clinical presentation with a Positive and Negative Syndrome Scale (PANSS) Total Score ≥ 80 AND
  * Specific psychotic symptoms on the PANSS as measured by a score of > 4 on each of the following items (possible scores of 1 to 7 for each item)

    * Conceptual disorganization (P2)
    * Hallucinatory behavior (P3)
    * Suspiciousness/persecution (P6)
    * Unusual thought content (G9)
* Subjects who have received previous outpatient antipsychotic treatment at an adequate dose for an adequate duration and who showed a previous good response to such antipsychotic treatment (other than clozapine) in last 12 months.
* Subjects with a history of relapse and/or exacerbation of symptoms when not receiving antipsychotic treatment, excluding current episode.
* Subjects willing to discontinue all prohibited psychotropic medications to meet protocol required washouts prior to and during trial period.
* BMI less ≤ 40 kg/m2 (morbid obesity) at screening.
* Subjects who are able to provide written informed consent.
* Ability to understand the nature of trial and follow protocol requirements.

Exclusion Criteria:

* Sexually active males of childbearing potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 180 days after last dose of trial medication. Sexually active females of childbearing potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 150 days after last dose of trial medication.
* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving IMP in this trial.
* Subjects with improvement of ≥ 30% in total PANSS score between the screening and baseline assessments. - Subjects presenting with a first episode of schizophrenia - Subjects hospitalized for ≥ 30 days out of the last 90 days prior to screening visit. Subjects who have been hospitalized > 5 days for current acute episode at the time of screening visit
* Subjects with schizophrenia who are considered resistant/refractory to antipsychotic treatment Subjects who have a history of response to clozapine treatment only.
* Subjects with a current DSM-IV-TR Axis I diagnosis other than schizophrenia Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder or mental retardation.
* Subjects experiencing acute depressive symptoms within past 30 days that require treatment with an antidepressant.
* Subjects with a significant risk of violent behavior; who represent a risk of committing suicide as indicated by any suicidal ideation within the last 1 month or any suicidal behaviors within the last year; or who present a serious risk of suicide.
* Subjects with clinically significant tardive dyskinesia,.
* Subjects with severe akathisia.
* Subjects who have met DSM-IV-TR criteria for substance abuse with past 3 months prior to screening or dependence within past 6 months; including alcohol and benzodiazepines, but excluding caffeine and nicotine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (35):
  - Little Rock, Arkansas
  - Springdale, Arkansas
  - Anaheim, California
  - Carson, California
  - Escondido, California
  - Long Beach, California
  - National City, California
  - Oakland, California
  - Oceanside, California
  - Pico Rivera, California
  - San Diego, California
  - Santa Ana, California
  - Sherman Oaks, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Kissimmee, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Hoffman Estates, Illinois
  - Lake Charles, Louisiana
  - Flowood, Mississippi
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Marlton, New Jersey
  - Holliswood, New York
  - Dayton, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
- Croatia (2):
  - Popovača
  - Zagreb
- Latvia (4):
  - Daugavpils
  - Jelgava
  - Liepāja
  - Strenči

REFERENCES:
- [Derived] Kane JM, Peters-Strickland T, Baker RA, Hertel P, Eramo A, Jin N, Perry PP, Gara M, McQuade RD, Carson WH, Sanchez R. Aripiprazole once-monthly in the acute treatment of schizophrenia: findings from a 12-week, randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2014 Nov;75(11):1254-60. doi: 10.4088/JCP.14m09168. PMID 25188501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was a Phase 3, multicenter, randomized, double-blind, placebo-controlled trial to assess the efficacy and safety of aripiprazole IM (intramuscular) depot as treatment for an acute episode of schizophrenia in adult participants. The trial was conducted in 55 sites.
Pre-assignment Details: This trial included a 13-Day Screening phase (which includes Washout from previous antipsychotics for 7 days and/or washout from other prohibited medications), a 12-Week acute treatment phase, and a 14 (±2) Day safety follow-up.
Groups:
- Aripiprazole IM Depot 400/300mg: Participants randomized to aripiprazole IM depot received aripiprazole IM depot 400 mg as the initial dose with a single decrease to aripiprazole IM depot 300 mg permitted for tolerability per the study physician. The study treatment was injected into gluteal muscle every 4 weeks (Baseline/Day, Week 4, Week 8) during the 12-Week Acute Treatment Phase (ie, 3 IM depot injections). For 14 days beginning with the first injection, participants received concomitant oral aripiprazole (10 to 20 mg/day based on the study physician's clinical judgment).
- Placebo: Participants randomized to Placebo group received matching placebo. For 14 days beginning with the first injection, participants received concomitant oral placebo.
Period: Overall Study
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo
Started | 168 | 172
Completed | 94 | 65
Not Completed | 74 | 107
Not completed — Lost to Follow-up | 9 | 10
Not completed — Adverse Event | 7 | 13
Not completed — Met Withdrawal Criteria | 7 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 35 | 17
Not completed — Lack of Efficacy | 15 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo | Total
Number analyzed (Participants) | 168 | 172 | 340
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.1 (11.0) | 42.7 (10.9) | 42.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 71
  Male | 130 | 139 | 269

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Endpoint in Positive and Negative Syndrome Scale (PANSS) Total Score.
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 that indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. The PANSS total score was the sum of the rating scores for 7 positive subscale items, 7 negative subscale items, and 16 general psychopathology subscale items from the PANSS panel. PANSS Total Score ranged from 30 (best possible outcome) to 210 (worst possible outcome). The primary statistical comparison was performed using the Mixed Model Repeated Measure (MMRM) approach.
Time Frame: Baseline to Week 10
Population: Efficacy sample was defined as the intent to treat (ITT) population which included randomized participants who took at least one injection of double-blind (aripiprazole IM depot or placebo) and had at least one Post-Baseline efficacy assessment. Data of only 162 and 167 participants from aripiprazole and placebo groups were available.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo
Number analyzed (Participants) | 162 | 167
Units on a scale
  Week 1 (N= 162, 167) | -8.9 (0.9) | -5.0 (0.9)
  Week 2 (N= 144, 157) | -15.2 (1.2) | -8.3 (1.2)
  Week 4 (N= 134, 140) | -19.0 (1.4) | -9.8 (1.3)
  Week 6 (N= 126, 117) | -21.5 (1.5) | -10.3 (1.5)
  Week 8 (N= 108, 96) | -23.7 (1.6) | -9.7 (1.6)
  Week 10 (N= 99, 81) | -26.8 (1.6) | -11.7 (1.6)
Statistical Analysis 1: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; Null hypothesis of change from Baseline in PANSS total score of aripiprazole IM depot 400/300mg group is same as that of placebo group was tested. The sample size estimated a 1:1 randomization ratio (aripiprazole IM depot 400/300mg: placebo) to achieve 90% power and to preserve a nominal alpha level of 0.05 given a treatment difference of -7.5 points in change from Baseline with standard deviation of 20 points between aripiprazole and placebo using a two-sided z-test; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — Kenward-Rodger degree of freedom was used to test the treatment effects and p-value was not adjusted as this is a primary efficacy endpoint; MMRM analysis with treatment, pooled centers, Week and treatment-by-Week, and Baseline-by-Week interaction as an unstructured covariate was performed; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-6.1 to -1.7] — Difference in Least Square (LS) mean of change and 95% Confidence interval were derived from pair-wise comparison within MMRM at Week 1
Statistical Analysis 2: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-10.0 to -4.0] — Difference in Least Square (LS) mean of change and 95% Confidence interval were derived from pair-wise comparison within MMRM at Week 2
Statistical Analysis 3: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.2, 95% CI 2-sided [-12.8 to -5.6] — Difference in Least Square (LS) mean of change and 95% Confidence interval were derived from pair-wise comparison within MMRM at week 4
Statistical Analysis 4: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.1, 95% CI 2-sided [-15.0 to -7.3] — Difference in Least Square (LS) mean of change and 95% Confidence interval were derived from pair-wise comparison within MMRM at Week 6
Statistical Analysis 5: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -14.0, 95% CI 2-sided [-18.4 to -9.6] — Difference in Least Square (LS) mean of change and 95% Confidence interval were derived from pair-wise comparison within MMRM at Week 8
Statistical Analysis 6: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -15.1, 95% CI 2-sided [-19.4 to -10.8] — Difference in Least Square (LS) mean of change and 95% Confidence interval were derived from pair-wise comparison within MMRM at Week 10

2. Secondary Outcome: Mean Change From Baseline to Endpoint in Clinical Global Impression-Severity Scale (CGI-S) Score.
Description: The severity of illness for each participants were rated using the CGI-S scale. The study physician were to answer the following question: "Considering your total experience with this particular population, how mentally ill is the patient at this time?" Response choices included were: 0= not assessed; 1= normal; not at all ill; 2= borderline mentally ill; 3= mildly ill; 4= moderately ill; 5= markedly ill; 6= severely ill; and 7= among the most extremely ill participants.
Time Frame: Baseline to Week 10
Population: Efficacy sample was defined as the intent to treat (ITT) population which included randomized participants who took at least one injection of double-blind (aripiprazole IM depot or placebo) and had at least one Post-Baseline efficacy assessment. Data of only 162 and 168 participants from aripiprazole and placebo groups were available.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo
Number analyzed (Participants) | 162 | 168
Units on a scale
  Week 1 (N= 162, 168) | -0.4 (0.1) | -0.2 (0.1)
  Week 2 (N= 144, 157) | -0.8 (0.1) | -0.4 (0.1)
  Week 4 (N= 134, 140) | -1.0 (0.1) | -0.4 (0.1)
  Week 6 (N= 126, 117) | -1.2 (0.1) | -0.5 (0.1)
  Week 8 (N= 108, 96) | -1.3 (0.1) | -0.6 (0.1)
  Week 10 (N= 99, 81) | -1.4 (0.1) | -0.6 (0.1)
Statistical Analysis 1: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; Null hypothesis of change from Baseline in PANSS total score of aripiprazole IM depot 400/300mg group is same as that of placebo group was tested; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — After the comparison for primary efficacy endpoint was statistically significant, the comparison of change from Baseline in CGI severity score was conducted at same alpha level 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.4 to -0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.7 to -0.4] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-0.9 to -0.5] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-0.9 to -0.5] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.1 to -0.6] — [estimate comment as in outcome 1, analysis 6]

3. Secondary Outcome: Mean Change From Baseline to Endpoint in PANSS Positive Subscale Score.
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. In positive subscale, the 7 positive symptom constructs were: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. PANSS Positive Subscale Score ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline to Week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo
Number analyzed (Participants) | 162 | 167
Units on a scale
  Week 1 (N= 162, 167) | -3.5 (0.3) | -2.1 (0.3)
  Week 2 (N= 144, 157) | -5.7 (0.4) | -3.4 (0.4)
  Week 4 (N= 134, 140) | -7.0 (0.5) | -3.9 (0.4)
  Week 6 (N= 126, 117) | -8.2 (0.5) | -4.4 (0.5)
  Week 8 (N= 108, 96) | -8.9 (0.5) | -4.1 (0.5)
  Week 10 (N= 99, 81) | -10.0 (0.5) | -4.9 (0.5)
Statistical Analysis 1: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.1 to -0.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-3.3 to -1.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-4.3 to -2.0] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-5.1 to -2.6] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-6.2 to -3.4] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-6.4 to -3.7] — [estimate comment as in outcome 1, analysis 6]

4. Secondary Outcome: Mean Change From Baseline to Endpoint in PANSS Negative Subscale Score.
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicated- absence of symptoms and a score of 7 indicated- extremely severe symptoms. The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs were: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation and stereotyped thinking. PANSS Negative Subscale Score ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline to Week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo
Number analyzed (Participants) | 162 | 167
Units on a scale
  Week 1 (N= 162, 167) | -1.6 (0.2) | -0.7 (0.2)
  Week 2 (N= 144, 157) | -2.4 (0.3) | -1.2 (0.3)
  Week 4 (N= 134, 140) | -3.1 (0.4) | -1.3 (0.4)
  Week 6 (N= 126, 117) | -3.5 (0.4) | -1.3 (0.4)
  Week 8 (N= 108, 96) | -4.0 (0.4) | -1.4 (0.4)
  Week 10 (N= 99, 81) | -4.5 (0.5) | -1.6 (0.5)
Statistical Analysis 1: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.6 to -0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0032, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.0 to -0.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-2.7 to -0.8] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.2 to -1.3] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-3.7 to -1.4] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-4.1 to -1.6] — [estimate comment as in outcome 1, analysis 6]

5. Secondary Outcome: Mean Change From Baseline to Endpoint in Personal and Social Performance Scale (PSP) Score.
Description: The PSP was a validated clinician scale that measured personal and social functionining in 4 domains: socially useful activities eg, work and study), personal and social relationships, self-care, disturbing and aggressive behaviours. Impairement in each of these domains was rated as absent, mild, manifest, marked, severe, or very severe. These ratings were then converted to a total score based on a 100-point scale using algorithms to identify the appropriate 10-point interval and the study physician's judgement to determine the total score within the 10-point interval. Participants with a PSP total score of 71 to 100 were considered to have mild functional difficulty. Scores of 31 to 70 represented varying degrees of disability (31 to 70) and ratings of 1 to 30 indicated minimal functioning that required intense support and/or supervision.
Time Frame: Week 10
Population: Efficacy sample included participants who took at least one injection of double-blind (aripiprazole IM depot or placebo) and had one Post-Baseline efficacy assessment. LOCF was used to impute the missing data with the recorded value obtained at the preceding visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo
Number analyzed (Participants) | 139 | 146
Units on a scale | 12.3 (1.2) | 5.2 (1.2)
Statistical Analysis 1: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; Statistical analysis for Week 10; Test type: Superiority or Other; p < .0001, ANCOVA; ANCOVA model with treatment and pooled centers as factors and Baseline value as covariate for the comparison at other visits; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [4.1 to 10.1] — Difference in least square mean of change were derived from ANCOVA model

6. Secondary Outcome: Mean Clinical Global Impression-Improvement Scale (CGI-I) Score at Endpoint.
Description: as for outcome 2
Time Frame: Week 10
Population: Efficacy sample was defined as the ITT population which included randomized participants who took at least one injection of double-blind (aripiprazole IM depot or placebo) and had at least one Post-Baseline efficacy assessment. LOCF was used to impute the missing data with the recorded value obtained at the preceding visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo
Number analyzed (Participants) | 162 | 168
Units on a scale | 2.7 (1.2) | 3.7 (1.3)
Statistical Analysis 1: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; Statistical analysis for Week 10. LOCF method were used in imputation of missing data; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; CMH raw mean scores differ test (Van Elteren test) controlling for pooled centers

7. Secondary Outcome: Responder Rate Based on PANSS Total Score.
Description: Responder rate was defined as ≥30% reduction from Baseline in PANSS Total Score. PANSS Total Score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Week 10
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo
Number analyzed (Participants) | 162 | 168
participants | 60 | 24
Statistical Analysis 1: Comparison: Aripiprazole IM Depot 400/300mg vs Placebo; Statistical analysis for Week 10. LOCF method were used in imputation of missing data; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; CMH test controlling by region (pooled sites); Mean Difference (Final Values) = 22.7, 95% CI 2-sided [12.9 to 32.4]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from ICF signed untill Follow-up 14 (± 2) days.
Description: One participant was randomly assigned to aripiprazole IM depot 400 mg/ 300 mg, but was not treated and did not have any post-randomization assessments and was not included in safety or efficacy assessments.
Arm/Group | Aripiprazole IM Depot 400/300mg | Placebo
Serious Adverse Events (participants affected / at risk) | 8/167 | 6/172
Other Adverse Events (participants affected / at risk) | 91/167 | 68/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IM Depot 400/300mg (N=167) | Placebo (N=172)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 2
Schizophrenia (Psychiatric disorders) | 3 | 3
Substance abuse (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IM Depot 400/300mg (N=167) | Placebo (N=172)
Constipation (Gastrointestinal disorders) | 16 | 12
Dyspepsia (Gastrointestinal disorders) | 10 | 11
Toothache (Gastrointestinal disorders) | 9 | 8
Injection site pain (General disorders) | 9 | 1
Weight increased (Investigations) | 28 | 12
Akathisia (Nervous system disorders) | 19 | 6
Headache (Nervous system disorders) | 24 | 28
Sedation (Nervous system disorders) | 9 | 2
Agitation (Psychiatric disorders) | 9 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No